CLINICAL TRIAL: NCT04069598
Title: Statin Intolerance in Patients With Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: A-HIT 4-SI Study
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Statin Adverse Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Statin intolerance test — Statin intolerance test

SUMMARY:
Patients with acute coronary syndrome (MI, NSTEMI, USAP) will be included. They will be screened for statin intolernace for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome

Exclusion Criteria:

* Being on statin, having statin related side effects

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-03-02 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Statin intolerance | 6 months
  Number (percentage) of patients with statin intolerance

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Haseki, Istanbul
  - Siyami Ersek, Istanbul
  - Tepecik, Izmir
  - Ozcan Basaran, Muğla